CLINICAL TRIAL: NCT06252779
Title: Study on the Therapeutic Effect and Mechanism of Transcranial Plasma Stimulation in the Treatment of Chronic Insomnia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qinying Ma (Other)
Responsible Party: Sponsor-Investigator, Qinying Ma, chief physician, The First Hospital of Hebei Medical University
Organization: The First Hospital of Hebei Medical University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20221117
Record Dates: First submitted 2024-01-19; First posted 2024-02-12 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-02

CONDITIONS: Chronic Insomnia Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plasma stimulation therapy group (Experimental)
  Interventions: Device: Plasma therapy equipment
- False stimulation treatment group (Placebo Comparator)
  Interventions: Device: Fake therapeutic device

INTERVENTIONS:
Device: Plasma therapy equipment — The host of this product contains a high-voltage generator that can generate high-voltage electrical energy and deliver it to the treatment head. The air supply mechanism sends air to the ionization chamber inside the treatment head, which is ionized under the action of high-voltage electricity to generate thermal plasma, forming a particle flow mainly composed of active nitric oxide (pNO), which is then sprayed out from the nozzle of the treatment head to the target tissue of the human body. PNO particles can alter skin permeability, allowing them to act on specific parts of the body after transdermal absorption on the surface of the body.The patient will receive 14 days of treatment, with 20 minutes per day.
  Arms: Plasma stimulation therapy group
Device: Fake therapeutic device — False stimuli with the same appearance and pattern as Plasma therapy equipment.The patient will receive 14 days of treatment, with 20 minutes per day.
  Arms: False stimulation treatment group

SUMMARY:
This study is a single center study, led by Dr. Ma Qinying from the Department of Neurology at the First Hospital of Hebei Medical University. This study is an intervention study on plasma stimulation, involving patients with insomnia disorders to observe the effectiveness of plasma stimulation on insomnia disorders. Collect the Hamilton Anxiety Scale, Hamilton Depression Scale, Pittsburgh Sleep Quality Index Scale, Insomnia Severity Index Scale, and Somatization Symptom Self Rating Scale from patients before and after intervention. Transcranial magnetic stimulation synchronous electroencephalogram (TMS-EEG) and functional magnetic resonance imaging data. The research period is from December 2023 to July 2025, and a total of 40 patients are planned to be included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, gender is not limited;
2. right-handed;
3. the audiovisual level is sufficient to complete the examinations required for the study;
4. No medication for 1 month before enrollment, or stable taking sleep-improving drugs but poor treatment effect;
5. Informed consent signed by the patient or family member.

Exclusion Criteria:

1. Substance abuse/dependence within 6 months prior to enrollment;
2. Have had other mental illnesses within 6 months prior to enrollment;
3. Those with severe or unstable organic diseases;
4. pregnant or lactating women;
5. Those with a score of 3 (suicide) in 17 items of the Hamilton Depression Rating Scale ≥ 3;
6. Those who have participated in any other clinical trials within 1 month before enrollment;
7. In the opinion of the investigator, there is a situation that is not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Functional magnetic resonance imaging | Before and after 14 day/false stimulation, 20 minutes each time
  Functional magnetic resonance imaging (fMRI) is an imaging technique based on blood oxygen level dependence (BOLD), which can display small changes in magnetic resonance signals caused by changes in blood oxygenation status in venous capillaries in various regions of the brain.
Transcranial Magnetic Stimulation Combined Electroencephalography | Before and after 14 day/false stimulation, 20 minutes each time
  with the advancement of technology, magnetic compatible EEG electrodes and amplifiers have been invented, making it possible to synchronously record undisturbed EEG under transcranial magnetic stimulation. The monitoring technology of transcranial magnetic stimulation combined electroencephalography (TMS-EEG) has also emerged

SECONDARY OUTCOMES:
Insomnia Severity Index Scale | Follow up for 10 minutes before and after 14 days of false stimulation, as well as one month after the completion of true/false stimulation
  ISI includes 7 questions that assess the severity and impact of insomnia, as well as its impact on daily function and psychological state.
Pittsburgh Sleep Quality Index Scale | Follow up for 10 minutes before and after 14 days of false stimulation, as well as one month after the completion of true/false stimulation
  PSQI was developed by Pittsburgh psychiatrist Buysse in the United States to evaluate the sleep quality of participants in the past month. It is suitable for evaluating the sleep quality of patients with sleep disorders and mental disorders, as well as for evaluating the sleep quality of the general population
Hamilton Anxiety Scale | Follow up for 10 minutes before and after 14 days of false stimulation, as well as one month after the completion of true/false stimulation
  Neurological examination scale for evaluating the anxiety status of subjects in the past month
Hamilton Depression Scale | Follow up for 10 minutes before and after 14 days of false stimulation, as well as one month after the completion of true/false stimulation
  Neurological examination scale for evaluating the depression status of subjects in the past month
Somatization Symptom Self Rating Scale | Follow up for 10 minutes before and after 14 days of false stimulation, as well as one month after the completion of true/false stimulation
  This scale can effectively assist non psychotherapists in identifying physical symptom disorders in a timely and early manner

CONTACTS AND LOCATIONS:
Locations (1):
- Qinying Ma, Shijiazhuang, China